CLINICAL TRIAL: NCT01299610
Title: A Randomised, Double-blind, Placebo-controlled Study of Topical GW870086X Formulation in Subjects With Moderate or Severe Atopic Dermatitis
Brief Title: A Study to Test the Effect of 2 Different Doses of Topical GW870086X on Atopic Dermatitis Also Including a Postive Control and a Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 113434
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-05

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic Dermatitis; GW870086X; TIS; IGA
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GW870086 2.0% & 0.2% (Experimental): GW870086 2.0%, GW870086 0.2% & Placebo each applied to a separate specific lesion for 21±2 days.
  Interventions: Drug: GW870086 2.0%; Drug: GW870086 0.2%; Drug: Placebo
- GW870086 2.0% & FP 0.05% (Experimental): GW870086 2.0%, FP 0.05% & Placebo each applied to a separate specific lesion for 21±2 days.
  Interventions: Drug: GW870086 2.0%; Drug: FP 0.05%; Drug: Placebo
- GW870086 0.2% & FP 0.05% (Experimental): GW870086 0.2%, FP 0.05% & Placebo each applied to a separate specific lesion for 21±2 days.
  Interventions: Drug: GW870086 0.2%; Drug: FP 0.05%; Drug: Placebo

INTERVENTIONS:
Drug: GW870086 2.0% — White to slightly colored opaque cream
  Arms: GW870086 2.0% & FP 0.05%; GW870086 2.0% & 0.2%
Drug: GW870086 0.2% — White to slightly colored opaque cream
  Arms: GW870086 0.2% & FP 0.05%; GW870086 2.0% & 0.2%
Drug: FP 0.05% — White cream
  Arms: GW870086 0.2% & FP 0.05%; GW870086 2.0% & FP 0.05%
Drug: Placebo — White to slightly colored opaque cream

SUMMARY:
This study is a randomised, double-blind, placebo-controlled study to assess the efficacy of GW870086X cream formulation in subjects with moderate to severe atopic dermatitis. Subjects will be assigned to take 3 out of the 4 possible treatments for 21 ±2 days: GW870086X 0.2% cream, GW870086X 2% cream, FP 0.05% cream (as a positive control) and placebo cream. All subjects will be randomised to receive placebo cream. Three index lesions located on the arms and/or legs (one on each) will be identified per subject and each treatment will be applied to the same lesion.

DETAILED DESCRIPTION:
This study is a randomised, double-blind, placebo-controlled study to assess the efficacy of GW870086X cream formulation in subjects with moderate to severe atopic dermatitis. The primary objective of this study is to assess 3 lesions using the Three Item Severity (TIS) score. The secondary objectives are to assess safety and tolerability of GW870086X, assess individual lesions using the Investigators Global Assessment (IGA) and to assess the pharmacokinetics of 21 days dosing of GW870086X administered as a cream. Twenty-five (25) subjects with atopic dermatitis will be randomised to receive placebo and 2 of the following treatments: GW870086X 0.2%, GW870086X 2%, FP 0.05% and placebo. All subjects will receive placebo. Subjects will apply all 3 treatments once daily during the 21 day treatment period. Three index lesions located on the arms and/or legs (one on each) will be identified per subject and each treatment will be applied to the same lesion throughout the 21±2 day treatment period. Each index lesion should represent the most common lesions for each patient i.e. not the most or least severe lesions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of atopic dermatitis who are otherwise healthy.
* Male or female between 18 and 65 years of age inclusive.
* A female subject is eligible to participate if she is of:

  • Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the protocol contraception methods if they wish to continue their HRT during the study.
* Male subjects with female partners of child-bearing potential must agree to use one of the protocol contraception methods.
* BMI within the range 19.0 - 29.0 kg/m2 (inclusive).
* Subjects must have body surface area (BSA) disease involvement of >5% as assessed by the rule of nines method.
* Patients must be willing to refrain from current active therapy for at least 10 days prior to dosing,
* Capable of giving written informed consent.
* Single QTc, QTcB < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* AST and ALT < 2xULN; alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* The subject presents with any systemic disorder, active skin disease or subjects who present with scars, moles, tattoos, body piercings, sunburn in the test area which could interfere with the assessment of lesions at screening.
* The subject has atopic dermatitis restricted to the face, the feet or the hands only.
* The subject has a current complication of atopic dermatitis for which treatment with anti-infectives are indicated.
* History of recent (< 6 months) active or presence of current superficial skin infections of viral aetiology
* The subject has been diagnosed as having contact dermatitis in area of target lesions, seborrheic dermatitis and/or occupational eczema at predilection sites of atopic dermatitis.
* The subject has had topical or transdermal treatments on or near the intended site of application within 14 days prior to first application of study medication.
* The subject has had systemic treatment for atopic dermatitis within 28 days of the first dose of study medication.
* Foreseeable intensive UV exposure during the study. Subjects must not be exposed to direct sunlight or skin tanning devices for the duration of the study.
* The subject has used topical treatment with tar or any corticosteroid within 14 days of the first dose of study medication except topical 1% hydrocortisone which may be used twice daily in patients with severe disease who require step-down therapy during the wash-out period until 3 days prior to study start, after which the hydrocortisone must be discontinued.
* The subject has used topical treatment with buproprion within 14 days of the first dose of study medication.
* History of cutaneous photodisorder.
* History of allergy to steroids or components of test medications.
* History or presence of skin (other than atopic dermatitis), hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Subjects with a history of diaphoresis/excessive sweating not restricted to palms or face.
* A positive test for Hepatitis B or Hepatitis C antibody.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-12-01; Primary Completion 2011-03-01 (Actual); Study Completion 2011-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 113434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113434 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at one center in Germany between 13 December 2010 and 14 April 2011.
Pre-assignment Details: Twenty five participants were randomized and completed the study.
Groups:
- Treatment 1: GW870086, 2.0%, GW870086, 0.2% and Placebo: Participants applied GW870086 2.0% cream, GW870086 0.2% cream and placebo cream to a separate specific lesion located on the arms and/or legs (one lesion per limb), applying same study treatment to the same lesion every day for 21±2 days. For first three days of the study, participants applied their randomly assigned treatments at the same time of day during the clinic visits and the study personnel supervised to ensure that the correct application procedures were followed. A full explanation was given to each participant regarding the labeling of the pots, the use of disposable gloves, the volume of cream to be used for each single application and the size of the area of skin to be treated. Participants applied their study treatments under supervision at the clinic on Days 7, 14 and 21 to allow accurately timed pharmacokinetic blood sampling and assessment of local tolerability. The participants applied their treatments at home on Day 4 to 6, Day 8 to 13 and Day 15 to 20.
- Treatment 2: GW870086 2.0%, FP 0.05% and Placebo: Participants applied GW870086 2.0% cream, Fluticasone Propionate (FP) 0.05% cream and placebo cream to a separate specific lesion located on the arms and/or legs (one lesion per limb), applying same study treatment to the same lesion every day for 21±2 days. For first three days of the study, participants applied their randomly assigned treatments at the same time of day during the clinic visits and study personnel supervised to ensure that the correct application procedures were followed. A full explanation was given to each participant regarding the labeling of pots, use of disposable gloves, the volume of cream to be used for each single application and the size of the area of skin to be treated. Participants applied their study treatments under supervision at the clinic on Days 7, 14 and 21 to allow accurately timed pharmacokinetic blood sampling and assessment of local tolerability. Participants applied their treatments at home on Day 4 to 6, Day 8 to 13 and Day 15 to 20.
- Treatment 3: GW870086 0.2%, FP 0.05% and Placebo: Participants applied GW870086 0.2% cream, FP 0.05% cream and placebo cream to a separate specific lesion located on the arms and/or legs (one lesion per limb), applying same study treatment to the same lesion every day for 21±2 days. For first three days of the study, participants applied their randomly assigned treatments at the same time of day during the clinic visits and study personnel supervised to ensure that the correct application procedures were followed. A full explanation was given to each participant regarding the labeling of pots, use of disposable gloves, the volume of cream to be used for each single application and the size of the area of skin to be treated. Participants applied their study treatments under supervision at the clinic on Days 7, 14 and 21 to allow accurately timed pharmacokinetic blood sampling and assessment of local tolerability. Participants applied their treatments at home on Day 4 to 6, Day 8 to 13 and Day 15 to 20.
Period: Overall Study
Arm/Group | Treatment 1: GW870086, 2.0%, GW870086, 0.2% and Placebo | Treatment 2: GW870086 2.0%, FP 0.05% and Placebo | Treatment 3: GW870086 0.2%, FP 0.05% and Placebo
Started | 10 | 5 | 10
Completed | 10 | 5 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment 1: GW870086, 2.0%, GW870086, 0.2% and Placebo: Participants applied GW870086, 2.0% cream, GW870086, 0.2% cream and placebo cream to a separate specific lesion located on the arms and/or legs (one lesion per limb), applying same study treatment to the same lesion every day for 21±2 days. For first three days of the study, participants applied their randomly assigned treatments at the same time of day during the clinic visits and the study personnel supervised to ensure that the correct application procedures were followed. A full explanation was given to each participant regarding the labeling of the pots, the use of disposable gloves, the volume of cream to be used for each single application and the size of the area of skin to be treated. Participants applied their study treatments under supervision at the clinic on Days 7, 14 and 21 to allow accurately timed pharmacokinetic blood sampling and assessment of local tolerability. The participants applied their treatments at home on Day 4 to 6, Day 8 to 13 and Day 15 to 20.
- Treatment 2: GW870086 2.0%, FP 0.05% and Placebo: Participants applied GW870086, 2.0% cream, Fluticasone Propionate (FP) 0.05% cream and placebo cream to a separate specific lesion located on the arms and/or legs (one lesion per limb), applying same study treatment to the same lesion every day for 21±2 days. For first three days of the study, participants applied their randomly assigned treatments at the same time of day during the clinic visits and study personnel supervised to ensure that the correct application procedures were followed. A full explanation was given to each participant regarding the labeling of pots, use of disposable gloves, the volume of cream to be used for each single application and the size of the area of skin to be treated. Participants applied their study treatments under supervision at the clinic on Days 7, 14 and 21 to allow accurately timed pharmacokinetic blood sampling and assessment of local tolerability. Participants applied their treatments at home on Day 4 to 6, Day 8 to 13 and Day 15 to 20.
- Treatment 3: GW870086 0.2%, FP 0.05% and Placebo: Participants applied GW870086, 0.2% cream, FP, 0.05% cream and placebo cream to a separate specific lesion located on the arms and/or legs (one lesion per limb), applying same study treatment to the same lesion every day for 21±2 days. For first three days of the study, participants applied their randomly assigned treatments at the same time of day during the clinic visits and study personnel supervised to ensure that the correct application procedures were followed. A full explanation was given to each participant regarding the labeling of pots, use of disposable gloves, the volume of cream to be used for each single application and the size of the area of skin to be treated. Participants applied their study treatments under supervision at the clinic on Days 7, 14 and 21 to allow accurately timed pharmacokinetic blood sampling and assessment of local tolerability. Participants applied their treatments at home on Day 4 to 6, Day 8 to 13 and Day 15 to 20.
- Total: Total of all reporting groups
Arm/Group | Treatment 1: GW870086, 2.0%, GW870086, 0.2% and Placebo | Treatment 2: GW870086 2.0%, FP 0.05% and Placebo | Treatment 3: GW870086 0.2%, FP 0.05% and Placebo | Total
Number analyzed (Participants) | 10 | 5 | 10 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.9 (18.81) | 40.8 (19.43) | 28.3 (10.15) | 36.2 (16.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 6
  Male | 7 | 3 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 5 | 10 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Three Item Severity (TIS) Scores Between GW870086 (0.2% and 2%) Versus Placebo at Day 22
Description: Three target lesions were selected and each of the 3 target lesions were assessed separately using the TIS for erythema, oedema/papulation, and excoriation using a score of 0 - 3 as 0 = absent, 1 = mild, 2 = moderate, 3 = severe. Each participant had at least 3 index lesions (=> 1square centimeter in size) with a sum score of =>4 and =< 6 for erythema, oedema/populations and excoriations using the TIS rating scale at screening. The index lesions represented common lesions i.e. not the most or least severe lesions. The total TIS score for a lesion was calculated as the sum of each of the component scores i.e. ranging from 0 (no symptoms) to 9 (severe symptoms). The values of Day 1 assessments were considered as Baseline values. The change from Baseline was calculated by subtracting the Baseline TIS score from Day 22 TIS score.
Time Frame: Baseline (Day 1) and Day 22
Population: The Efficacy Population was defined as participants in the 'All Subjects' population with at least one post dose TIS assessment.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Groups:
- GW870086, 0.2% Cream: Participants applied GW870086, 0.2% cream to a specific lesion located on the arms and/or legs every day for 21±2 days. For first three days of the study, participants applied their randomly assigned treatments at the same time of day during the clinic visits and study personnel supervised to ensure that the correct application procedures were followed. A full explanation was given to each participant regarding the labeling of pots, use of disposable gloves, the volume of cream to be used for each single application and the size of the area of skin to be treated. Participants applied their study treatments under supervision at the clinic on Days 7, 14 and 21 to allow accurately timed pharmacokinetic blood sampling and assessment of local tolerability. Participants applied their treatments at home on Day 4 to 6, Day 8 to 13 and Day 15 to 20.
- GW870086, 2.0% Cream: Eligible participants applied GW870086, 2.0% cream to a specific lesion located on the arms and/or legs every day for 21±2 days. For first three days of the study, participants applied their randomly assigned treatments at the same time of day during the clinic visits and study personnel supervised to ensure that the correct application procedures were followed. A full explanation was given to each participant regarding the labeling of pots, use of disposable gloves, the volume of cream to be used for each single application and the size of the area of skin to be treated. Participants applied their study treatments under supervision at the clinic on Days 7, 14 and 21 to allow accurately timed pharmacokinetic blood sampling and assessment of local tolerability. Participants applied their treatments at home on Day 4 to 6, Day 8 to 13 and Day 15 to 20.
- Placebo: Eligible participants applied matching placebo to a specific lesion located on the arms and/or legs every day for 21±2 days. For first three days of the study, participants applied their randomly assigned treatments at the same time of day during the clinic visits and study personnel supervised to ensure that the correct application procedures were followed. A full explanation was given to each participant regarding the labeling of pots, use of disposable gloves, the volume of cream to be used for each single application and the size of the area of skin to be treated. Participants applied their study treatments under supervision at the clinic on Days 7, 14 and 21 to allow accurately timed pharmacokinetic blood sampling and assessment of local tolerability. Participants applied their treatments at home on Day 4 to 6, Day 8 to 13 and Day 15 to 20.
- FP, 0.05% Cream: Eligible participants applied FP, 0.05% cream to a specific lesion located on the arms and/or legs every day for 21±2 days. For first three days of the study, participants applied their randomly assigned treatments at the same time of day during the clinic visits and study personnel supervised to ensure that the correct application procedures were followed. A full explanation was given to each participant regarding the labeling of pots, use of disposable gloves, the volume of cream to be used for each single application and the size of the area of skin to be treated. Participants applied their study treatments under supervision at the clinic on Days 7, 14 and 21 to allow accurately timed pharmacokinetic blood sampling and assessment of local tolerability. Participants applied their treatments at home on Day 4 to 6, Day 8 to 13 and Day 15 to 20.
Arm/Group | GW870086, 0.2% Cream | GW870086, 2.0% Cream | Placebo | FP, 0.05% Cream
Number analyzed (Participants) | 20 | 15 | 25 | 15
Score on scale | -1.99 (0.418) | -2.49 (0.465) | -1.61 (0.380) | -3.11 (0.467)
Statistical Analysis 1: Comparison: GW870086, 0.2% Cream vs Placebo; Test type: Superiority or Other; p = 0.480, Mixed model for repeated measures; Difference in Adjusted Means = -0.38, 95% CI 2-sided [-1.46 to 0.70], Standard Error of Mean 0.538
Statistical Analysis 2: Comparison: GW870086, 2.0% Cream vs Placebo; Test type: Superiority or Other; p = 0.118, Mixed model for repeated measures; mixed model for repeated measures = -0.89, 95% CI 2-sided [-2.00 to 0.23], Standard Error of Mean 0.557
Statistical Analysis 3: Comparison: Placebo vs FP, 0.05% Cream; Test type: Superiority or Other; p = 0.011, Mixed model for repeated measures; Difference in Adjusted Means = -1.51, 95% CI 2-sided [-2.65 to -0.36], Standard Error of Mean 0.572

2. Secondary Outcome: Change From Baseline TIS Scores Between GW870086X (0.2% and 2%) Versus Placebo on Days 2, 3, 7 and 14
Description: Three target lesions were selected and each of the 3 target lesions were assessed separately using the TIS for erythema, oedema/papulation, and excoriation using a score of 0 - 3 as 0 = absent, 1 = mild, 2 = moderate, 3 = severe. Each participant had at least 3 index lesions (=> 1square centimeter in size) with a sum score of =>4 and =< 6 for erythema, oedema/populations and excoriations using the TIS rating scale at screening. The index lesions represented common lesions i.e. not the most or least severe lesions. The total TIS score for a lesion was calculated as the sum of each of the component scores i.e. may range from 0 (no symptoms) to 9 (severe symptoms). The values of Day 1 assessments were considered as Baseline values. The change from Baseline was calculated by subtracting the Baseline TIS score from Day 22 values TIS score.
Time Frame: Days 2, 3, 7, and 14
Population: Efficacy Population
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | GW870086, 0.2% Cream | GW870086, 2.0% Cream | Placebo | FP, 0.05% Cream
Number analyzed (Participants) | 20 | 15 | 25 | 15
Score on scale
  Day 2 | -0.37 (0.19) | -0.53 (0.203) | -0.45 (0.181) | -0.62 (0.203)
  Day 3 | -0.91 (0.266) | -0.80 (0.291) | -0.94 (0.246) | -1.22 (0.292)
  Day 7 | -1.43 (0.363) | -1.78 (0.403) | -1.19 (0.331) | -2.47 (0.405)
  Day 14 | -1.82 (0.367) | -2.23 (0.408) | -1.58 (0.335) | -2.97 (0.409)
Statistical Analysis 1: Comparison: GW870086, 0.2% Cream vs Placebo; GW870086, 0.2% cream Vs Placebo: Day 2; Test type: Superiority or Other; p = 0.581, Mixed model repeated measures; Difference in Adjusted Means = 0.09, 95% CI 2-sided [-0.24 to 0.42], Standard Error of Mean 0.160
Statistical Analysis 2: Comparison: GW870086, 2.0% Cream vs Placebo; GW870086, 2.0% cream Vs Placebo: Day 2; Test type: Superiority or Other; p = 0.655, Mixed model repeated measures; Difference in Adjusted Means = -0.08, 95% CI 2-sided [-0.42 to 0.27], Standard Error of Mean 0.169
Statistical Analysis 3: Comparison: Placebo vs FP, 0.05% Cream; FP, 0.05% cream Vs Placebo: Day 2; Test type: Superiority or Other; p = 0.336, Mixed model repeated measures; Difference in Adjusted Means = -0.17, 95% CI [-0.52 to 0.18], Standard Error of Mean 0.174
Statistical Analysis 4: Comparison: GW870086, 0.2% Cream vs Placebo; GW870086 0.2% cream Vs Placebo: Day 3; Test type: Superiority or Other; p = 0.923, Mixed model repeated measures; Difference in Adjusted Means = 0.03, 95% CI 2-sided [-0.58 to 0.63], Standard Error of Mean 0.302
Statistical Analysis 5: Comparison: GW870086, 2.0% Cream vs Placebo; GW870086, 2.0% cream, Placebo: Day 3; Test type: Superiority or Other; p = 0.657, Mixed model repeated measures; Difference in Adjusted Means = 0.14, 95% CI 2-sided [-0.49 to 0.77], Standard Error of Mean 0.314
Statistical Analysis 6: Comparison: Placebo vs FP, 0.05% Cream; Placebo, FP, 0.05% cream: Day 3; Test type: Superiority or Other; p = 0.386, Mixed model repeated measures; Difference in Adjusted Means = -0.28, 95% CI 2-sided [-0.93 to 0.36], Standard Error of Mean 0.323
Statistical Analysis 7: Comparison: GW870086, 0.2% Cream vs Placebo; GW870086, 0.2% cream, Placebo: Day 7; Test type: Superiority or Other; p = 0.601, Mixed model repeated measures; Difference in Adjusted Means = -0.24, 95% CI 2-sided [-1.15 to 0.67], Standard Error of Mean 0.456
Statistical Analysis 8: Comparison: GW870086, 2.0% Cream vs Placebo; GW870086, 2.0% cream, Placebo: Day 7; Test type: Superiority or Other; p = 0.212, Mixed model repeated measures; Difference in Adjusted Means = -0.60, 95% CI 2-sided [-1.54 to 0.35], Standard Error of Mean 0.472
Statistical Analysis 9: Comparison: Placebo vs FP, 0.05% Cream; Placebo, FP, 0.05% cream: Day 7; Test type: Superiority or Other; p = 0.010, Mixed model repeated measures; Difference in Adjusted Means = -1.29, 95% CI 2-sided [-2.26 to -0.32], Standard Error of Mean 0.485
Statistical Analysis 10: Comparison: GW870086, 0.2% Cream vs Placebo; GW870086, 0.2% cream, Placebo: Day 14; Test type: Superiority or Other; p = 0.602, Mixed model repeated measures; Difference in Adjusted Means = -0.24, 95% CI 2-sided [-1.17 to 0.68], Standard Error of Mean 0.462
Statistical Analysis 11: Comparison: GW870086, 2.0% Cream vs Placebo; GW870086, 2.0% cream, Placebo: Day 14; Test type: Superiority or Other; p = 0.180, Mixed model repeated measures; Difference in Adjusted Means = -0.65, 95% CI 2-sided [-1.61 to 0.31], Standard Error of Mean 0.479
Statistical Analysis 12: Comparison: Placebo vs FP, 0.05% Cream; Placebo, FP, 0.05% cream: Day 14; Test type: Superiority or Other; p = 0.006, Mixed model repeated measures; Difference in Adjusted Means = -1.39, 95% CI 2-sided [-2.37 to -0.40], Standard Error of Mean 0.492

3. Secondary Outcome: Number of Investigators Global Assessment (IGA) Responders on Days 2, 3, 7, 14 and 22
Description: Three target lesions were selected and each of the 3 target lesions were assessed separately using the IGA. The IGA was carried out by a trained dermatologist and score ranged from 0 to 5. The detailed IGA scale is as: 0-Clear: No inflammatory signs of atopic dermatitis, 1- Almost clear: Just perceptible erythema and just perceptible apulation/infiltration, 2-Mild: Mild erythema and mild papulation/infiltration, 3-Moderate: Moderate erythema, and moderate papulation/infiltration, 4-Severe: Severe erythema and severe papulation/infiltration, 5-Very Severe: Very severe erythema, and very severe papulation/infiltration with oozing/crusting. The participant was considered as responder if each lesion at timepoint, IGA score reduced by 1 grade and improved from Baseline by 2 grades.
Time Frame: Days 2, 3, 7, 14 and 22
Population: Efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | GW870086, 0.2% Cream | GW870086, 2.0% Cream | Placebo | FP, 0.05% Cream
Number analyzed (Participants) | 20 | 15 | 25 | 15
Participants
  Day 2 | 0 | 0 | 1 | 2
  Day 3 | 0 | 0 | 1 | 1
  Day 7 | 3 | 1 | 1 | 6
  Day 14 | 8 | 2 | 4 | 6
  Day 22 | 6 | 4 | 7 | 11

4. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE include AEs those result in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Number of participants with AEs and SAEs were reported.
Time Frame: Upto Day 21
Population: All Subjects Population was defined as all participants who had at least one application of placebo, GW870086X 0.2%, GW 870086X 2% or FP 0.05% cream.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: GW870086, 2.0%, GW870086, 0.2% and Placebo | Treatment 2: GW870086 2.0%, FP 0.05% and Placebo | Treatment 3: GW870086 0.2%, FP 0.05% and Placebo
Number analyzed (Participants) | 10 | 5 | 10
Participants
  Any AEs | 6 | 2 | 5
  Any SAEs | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Abnormal Hematology and Clinical Chemistry Parameters of Potential Clinical Importance (PCI)
Description: Laboratory ranges of PCI represented as multiplier of lower limit of normal [LLN]; Multipliers of upper limit of normal (ULN). Laboratory ranges of PCI for white blood cell count (0.67×LLN; 1.82×ULN), neutrophil count (0.83×ULN), hemoglobin for male (1.03×ULN) and for female (1.13×ULN), hematocrit for male (1.02×ULN) for female (1.17×ULN), platelet count (0.67×LLN; 1.57), lymphocytes (0.81×LLN), albumin (0.86 ×LLN), calcium (0.91×LLN; 1.06×ULN), glucose (0.71×LLN; 1.41×ULN), potassium (0.86×LLN; 1.10×ULN), sodium (0.96×LLN; 1.03×ULN), aspartate amino transferase (>= 2x ULN), alanine transaminase (>=2x ULN), alkaline Phosphatase (>=2x ULN), total bilirubin (>=1.5x ULN). Only those parameters for which at least one value of PCI was reported are summarized. The number of participants with PCI hematology and clinical chemistry findings at any visit during the treatment and follow-up were reported.
Time Frame: Up to Day 21
Population: All subject population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: GW870086, 2.0%, GW870086, 0.2% and Placebo | Treatment 2: GW870086 2.0%, FP 0.05% and Placebo | Treatment 3: GW870086 0.2%, FP 0.05% and Placebo
Number analyzed (Participants) | 10 | 5 | 10
Participants
  Lymphocyte, Low | 1 | 0 | 1
  Total Neutrophils, Low | 1 | 0 | 0
  AST, High | 0 | 0 | 1
  Glucose, Low | 0 | 0 | 1

6. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) of PCI
Description: 12-lead ECG was obtained. The standard ECG criteria of PCI were 1) absolute QTc Interval, > 450 milliseconds (msec), 2) increase from Baseline in QTc > 60 msec 3) absolute PR Interval, <110 and >220 msec, 4) absolute QRS Interval, < 75 and >110 msec. The number of participants with PCI ECG findings at any visit during the treatment and follow-up were reported.
Time Frame: Up to Day 21
Population: All subject population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: GW870086, 2.0%, GW870086, 0.2% and Placebo | Treatment 2: GW870086 2.0%, FP 0.05% and Placebo | Treatment 3: GW870086 0.2%, FP 0.05% and Placebo
Number analyzed (Participants) | 10 | 5 | 10
Participants | 1 | 1 | 1

7. Secondary Outcome: Number of Participants With Abnormal Vital Signs (Systolic and Diastolic Blood Pressure and Pulse Rate) of PCI
Description: The PCI ranges (low and high) of the vital sign parameters were for systolic blood pressure (<85 and >160 millimeter of mercury [mmHg]), diastolic blood pressure (<45 and >100 mmHg) and heart rate (<40 and >110 beats per minute). Only those parameters for which at least one value of PCI was reported are summarized. There were no values of PCI in vital signs parameters over the course of the study.
Time Frame: Up to Day 21
Population: All subject population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1: GW870086, 2.0%, GW870086, 0.2% and Placebo | Treatment 2: GW870086 2.0%, FP 0.05% and Placebo | Treatment 3: GW870086 0.2%, FP 0.05% and Placebo
Number analyzed (Participants) | 10 | 5 | 10
Participants | 0 | 0 | 0

8. Secondary Outcome: Pharmacokinetic Parameters: Maximum Observed Concentration (Cmax) of GW870086X
Description: Cmax was planned to be determined directly from the raw concentration-time data. The pharmacokinetic parameters were planned to be calculated by standard non-compartmental analysis using Win-Nonlin Pro-Version 5.2 or higher.
Time Frame: Day 7, 14 and 21
Population: Pharmacokinetic population was defined as participants in the All Subjects population for whom a pharmacokinetic sample was obtained and analyzed. Cmax was not analysed because the plasma concentrations were not quantifiable.
Arm/Group | GW870086, 0.2% Cream | GW870086, 2.0% Cream | Placebo | FP, 0.05% Cream
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Pharmacokinetic Parameter: Time of Occurrence of Cmax (Tmax) of GW870086
Description: Tmax was planned to be determined directly from the raw concentration-time data. The pharmacokinetic parameters were planned to be calculated by standard non-compartmental analysis using Win-Nonlin Pro-Version 5.2 or higher.
Time Frame: Day 7, 14 and 21
Population: Pharmacokinetics population. Tmax was not analysed because the plasma concentrations were not quantifiable.
Arm/Group | GW870086, 0.2% Cream | GW870086, 2.0% Cream | Placebo | FP, 0.05% Cream
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Pharmacokintics Parameter: Area Under Curve (AUC) of GW870086
Description: The area under the plasma concentration-time curve to the last quantifiable concentration (AUC[0-t]) and area under the plasma concentration-time curve over the dosing interval (AUC[0-tou]) was planned to be determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. The pharmacokinetic parameters were planned to be calculated by standard non-compartmental analysis using Win-Nonlin Pro-Version 5.2 or higher.
Time Frame: Day 7, 14 and 21
Population: Pharmacokinetics population. AUC was not analyzed because the plasma concentrations were not quantifiable.
Arm/Group | GW870086, 0.2% Cream | GW870086, 2.0% Cream | Placebo | FP, 0.05% Cream
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Pharmacodynamics Endpoint: Skin Thickness and Other Markers of Atopic Dermatitis
Description: A 4 millimeter (mm) punch skin biopsy was taken pre- and post-treatment (Day 1 and Day 21) from each of the 3 index lesions. The results were not analyzed for this outcome measure.
Time Frame: Day 1 and Day 22
Population: Efficacy Population
Arm/Group | GW870086, 0.2% Cream | GW870086, 2.0% Cream | Placebo | FP, 0.05% Cream
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from the start of study treatment (Day 1) and until the follow-up contact (approximately 7-14 days after last dose).
Description: All Subjects Population
Arm/Group | Treatment 1: GW870086, 2.0%, GW870086, 0.2% and Placebo | Treatment 2: GW870086 2.0%, FP 0.05% and Placebo | Treatment 3: GW870086 0.2%, FP 0.05% and Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 2/5 | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1: GW870086, 2.0%, GW870086, 0.2% and Placebo (N=10) | Treatment 2: GW870086 2.0%, FP 0.05% and Placebo (N=5) | Treatment 3: GW870086 0.2%, FP 0.05% and Placebo (N=10)
Headache (Nervous system disorders) | 2 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.